CLINICAL TRIAL: NCT00515476
Title: Randomized, Clinical Trial to Study the Effect of Exercise Training on the Function of HDL-Cholesterol, Endothelial Function, Oxidative Stress and Regenerative Capacity of Endothelial Progenitor Cells in Patients With Metabolic Syndrome
Brief Title: Effect of Exercise Training on the Function of the High Density Lipoprotein (HDL)-Cholesterol, Endothelial Function and Endothelial Progenitor Cells in Patients With Metabolic Syndrome(HERMET-Study)
Acronym: HERMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Pricipal Investigator Prof. Dr. med. H. Drexler, MHH Hannover Medical School
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4031215
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2009-11

CONDITIONS: Metabolic Syndrome X
Keywords: metabolic syndrome; HDL-Cholesterol; EPC; endothelial function; reduced blood HDL-Cholesterol level
MeSH Terms: conditions — Metabolic Syndrome | interventions — Exercise

INTERVENTIONS:
Behavioral: physical exercise — 8 weeks of regular exercise training

SUMMARY:
The purpose of the present study is to characterize the quality of HDL-Cholesterol in patients with metabolic syndrome and reduced blood HDL-Cholesterol levels and to examine the effect of exercise training on the vasculoprotective effects of HDL-Cholesterol in these patients. Additionally the investigators aim to investigate the endothelial function, oxidative stress and the regenerative capacity of the endothelial progenitor cells in patients with metabolic syndrome and the changes dependent on physical activity of patients.

ELIGIBILITY:
Inclusion Criteria:

* Reduced HDL-Cholesterol levels in blood: < 40 mg/dl (1.03 mmol/L) in male, < 50 mg/dl (1.29 mmol/L) in female
* Plus two of the following criteria:
* Elevated waist circumference: ≥ 102 cm (≥ 40 inches) in men or ≥ 88 cm (≥ 35 inches) in women
* Elevated triglycerides: ≥ 150 mg/dL (1.7 mmol/L
* Elevated blood pressure: ≥ 130 mmHg systolic blood pressure or ≥ 80 mmHg
* diastolic blood pressure or anti-hypertensive treatment
* Elevated fasting glucose: ≥ 100 mg/dL or on drug treatment for elevated fasting glucose

Exclusion Criteria:

* Acute coronary syndrome
* Unstable Angina pectoris
* Myocardial infarction during the last 8 weeks
* Therapy with Niacin
* Active infections
* Ventricular arrhythmias
* Systolic blood pressure > 160 mmHg or diastolic blood pressure > 95 mmHg
* Cancer
* Pregnancy, lactation
* Alcoholism

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Primary: vasculoprotective and regenerative functions of HDL-Cholesterol and EPC function before and after 8-weeks exercise training | before and after 8-weeks exercise training

SECONDARY OUTCOMES:
Secondary: flow-mediated, endothelium-dependent vasodilation of radial artery measured by ultrasound | before and 8 weeks after exercise training

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Drexler, MD, Study Director — Hannover Medical School; Kristina Sonnenschein, MD, Principal Investigator — Hannover Medical School; Ulf Landmesser, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany

REFERENCES:
- [Derived] Sonnenschein K, Horvath T, Mueller M, Markowski A, Siegmund T, Jacob C, Drexler H, Landmesser U. Exercise training improves in vivo endothelial repair capacity of early endothelial progenitor cells in subjects with metabolic syndrome. Eur J Cardiovasc Prev Rehabil. 2011 Jun;18(3):406-14. doi: 10.1177/1741826710389373. Epub 2011 Feb 11. PMID 21450652